CLINICAL TRIAL: NCT06101563
Title: Optimal Duration Between Drainage for Obstructing Renal or Ureteral Stones Associated With Infection and Ureteroscopic Lithotripsy: A Randomized Controlled Trial.
Brief Title: Duration Between Drainage and Ureteroscopic Lithotripsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed R EL-Nahas, Professor of Urology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2371
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Ureter Stone; Renal Stone; Ureteric Obstruction
Keywords: Ureteroscopy; Sepsis; infectious complications; ureteric calculi; Renal calculi
MeSH Terms: conditions — Ureterolithiasis; Nephrolithiasis; Ureteral Obstruction; Sepsis; Kidney Calculi

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early (Active Comparator): Patients will be managed by ureteroscopic lithotripsy 7 days after drainage.
  Interventions: Procedure: Early ureteroscopy
- Delayed (Active Comparator): Patients will be managed by ureteroscopic lithotripsy 14-21 days after drainage.
  Interventions: Procedure: Delayed Ureteroscopy

INTERVENTIONS:
Procedure: Early ureteroscopy — Patients will be managed by ureteroscopic lithotripsy 7 days after drainage.
  Arms: Early
Procedure: Delayed Ureteroscopy — Patients will be managed by ureteroscopic lithotripsy 14-21 days after drainage.
  Arms: Delayed

SUMMARY:
This study will be conducted to compare early (seven days) versus delayed (14-21 days) definitive ureteroscopic lithotripsy after initial drainage for obstructing ureteral or renal stones associated with infection.

DETAILED DESCRIPTION:
All the study participants will be monitored during the early post-operative period for post-operative pain and complications. The rate and grade of reported complications will be determined according to modified Dindo-Clavian grading system. After ensuring safe status for discharge, all patients will be reassessed at the outpatient department after 4 weeks by NCCT to assess stone free status.

ELIGIBILITY:
Inclusion Criteria:

1. Obstructing ureteral or renal stone <20 mm.
2. Associated clinical evidence of acute upper urinary tract infection based on systemic inflammatory response syndrome (SIRS).

Exclusion Criteria:

1. History of endoscopic instrumentation to the urinary tract in the last 4 weeks prior to presentation.
2. Bilateral obstructed kidneys necessitating bilateral drainage.
3. Associated emphysematous pyelonephritis or perinephric abscess.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Percentage of postoperative infectious complications in treatment groups | 30 days
  Difference in post-URS infectious complications between the study groups. infectious complications are defined as presence of urinary tract infection with one of the following findings: - Body temperature more than 38.3C or below 36C. - Tachycardia (>90/minute). - Respiratory rate more than 20/minute. - Disturbed mental status. - Systolic blood pressure < 90 mmHg & mean arterial pressure < 70 mmHg or systolic blood pressure decrease < 40 mmHg. - WBC >12,000 or <4,000.

CONTACTS AND LOCATIONS:
Overall Officials: Yaser Osman, MD, Study Chair — Professor; Mahmoud Laymon, MD,MRCS, Study Chair — Lecturer
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No